CLINICAL TRIAL: NCT04614064
Title: Exposure to Particulate Matter on the London Underground in Healthy Subjects and Patients With Chronic Respiratory Disease
Brief Title: London Underground Study - Health Effects of Particulate Matter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 20SM6236
Record Dates: First submitted 2020-10-22; First posted 2020-11-03 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Chronic Obstructive Pulmonary Disease; Particulate matter; London Underground
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COPD patients (Experimental): As per inclusion and exclusion criteria for COPD patients
  Interventions: Other: Exposure to London Underground ambient particulate matter; Other: Exposure to London air ambient particulate matter
- Healthy volunteers (Experimental): As per inclusion and exclusion criteria for healthy volunteers
  Interventions: Other: Exposure to London Underground ambient particulate matter; Other: Exposure to London air ambient particulate matter

INTERVENTIONS:
Other: Exposure to London Underground ambient particulate matter — Exposure to particulate matter on the London Underground
Other: Exposure to London air ambient particulate matter — Exposure to ambient particulate matter on the London Overground (as a proxy as a proxy for a clean air London area while maintaining other aspects of a train journey)

SUMMARY:
An average of 4.8 million journeys are made on the London Underground every day and as the 'Tube' has elevated airborne particulate matter concentrations compared to ambient air, this raises concern about the potential health impact of this environment. This study explores the health effects of particulate matter from the London Underground on patients with COPD and healthy volunteers.

Patients with COPD and healthy participants will be invited to undertake a set 90 min journey on the London Underground, and on a separate occasion (3-8 weeks apart), a 90 min journey on the London Overground (as a proxy for a clean air London area while maintaining other aspects of a train journey). A series of clinical, physiological and inflammatory data will be collected before, during and after (at different time points) each of the sessions in order to compare their response in relation to exposure and/or to disease status.

ELIGIBILITY:
Inclusion Criteria for both groups:

* Give informed consent
* London resident

For participants with COPD:

* GOLD stage 2 COPD (FEV1/FVC<70%; 50%>FEV1<80% predicted), GOLD stage 3 COPD (FEV1/FVC<70%; 30%>FEV1<50%) and GOLD stage 4 (FEV1/FVC<70%;FEV1<30%)
* No history of ischaemic heart disease

For healthy volunteers:

* No history of ischaemic heart disease.
* Normal lung function with no evidence of airflow obstruction.

Exclusion Criteria for both participants with COPD and healthy volunteers:

* Those with unstable ischaemic heart disease or COPD.
* Current smokers and those who are ex-smokers of <12 months duration.
* Those who work in the London Underground or are occupationally exposed to - - high levels of vehicle traffic exposure on a frequent basis.
* Those who cannot walk for 30 mins.
* Involvement in another research study
* Those unable to give consent.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
The difference (London Underground vs control exposure) in post exposure pulse wave velocity in healthy vs COPD participants. | -2 hours, +2 hours, +5 hours, +6 hours, +24 hours
  Measurement of arterial stiffness

SECONDARY OUTCOMES:
Other clinical responses on the London Underground vs control exposure | -2 hours, 0 hours, +45 minutes +90 minutes, +4 hours, +5 hours, +6 hours, +24 hours
  Symptom questionnaire
Other clinical responses on the London Underground vs control exposure | -2 hours, 0 hours, +45 minutes, +90 minutes, +2 hours, +4 hours, +6 hours, +24 hours
  Spirometry (FEV1)
Other clinical responses on the London Underground vs control exposure | -2 hours, 0 hours, +45 minutes, +90 minutes, +2 hours, +4 hours, +6 hours, +24 hours
  Spirometry (FVC)
Other clinical responses on the London Underground vs control exposure | -2 hours, 0 hours, +45 minutes, +90 minutes, +2 hours, +4 hours, +6 hours, +24 hours
  Spirometry (FEF 25-75)
Other clinical responses on the London Underground vs control exposure | -2 hours, +7 hours, +24 hours
  Single breath transfer factor for carbon monoxide (TLCO)
Circulating inflammatory and oxidative responses after the exposure on the London Underground vs control exposure | -2 hours, +7 hours, +24 hours
  Blood sample (IL8)
Circulating inflammatory and oxidative responses after the exposure on the London Underground vs control exposure | -2 hours, +7 hours, +24 hours
  Blood sample (High sensitivity CRP)
Circulating inflammatory and oxidative responses after the exposure on the London Underground vs control exposure | -2 hours, +7 hours, +24 hours
  Blood sample (FBC)
Circulating inflammatory and oxidative responses after the exposure on the London Underground vs control exposure | -2 hours, +7 hours, +24 hours
  Blood sample (TNFa)
Circulating inflammatory and oxidative responses after the exposure on the London Underground vs control exposure | -2 hours, +7 hours, +24 hours
  Blood sample (vWf antigen)
Circulating inflammatory and oxidative responses after the exposure on the London Underground vs control exposure | -2 hours, +7 hours, +24 hours
  Blood sample (Thrombin generation (systemic inflammatory response))
Circulating inflammatory and oxidative responses after the exposure on the London Underground vs control exposure | -2 hours, +7 hours, +24 hours
  Blood sample (8-isoprostanes (ELISA))
Circulating inflammatory and oxidative responses after the exposure on the London Underground vs control exposure | -2 hours, +7 hours, +24 hours
  Blood sample (Blood malondialdehyde (lipid peroxidation))
Circulating inflammatory and oxidative responses after the exposure on the London Underground vs control exposure | -2 hours, +7 hours, +24 hours
  Blood sample (Oxidation Reduction Potential (oxidative stress))
Circulating inflammatory and oxidative responses after the exposure on the London Underground vs control exposure | -2 hours, +7 hours, +24 hours
  Nasosorption (IL-8)
Circulating inflammatory and oxidative responses after the exposure on the London Underground vs control exposure | -2 hours, +7 hours, +24 hours
  Nasosorption (IL-6)
Circulating inflammatory and oxidative responses after the exposure on the London Underground vs control exposure | -2 hours, +7 hours, +24 hours
  Nasosorption (IL-33)
Circulating inflammatory and oxidative responses after the exposure on the London Underground vs control exposure | -2 hours, +7 hours, +24 hours
  Nasosorption (Myeloperoxidase)
Circulating inflammatory and oxidative responses after the exposure on the London Underground vs control exposure | -2 hours, +7 hours, +24 hours
  Nasosorption (Neutrophil lipocalin-2)
Circulating inflammatory and oxidative responses after the exposure on the London Underground vs control exposure | -2 hours, +7 hours, +24 hours
  Nasosorption (Tryptases)
Circulating inflammatory and oxidative responses after the exposure on the London Underground vs control exposure | -2 hours, +7 hours, +24 hours
  Nasosorption (Complement)
Circulating inflammatory and oxidative responses after the exposure on the London Underground vs control exposure | -2 hours, +7 hours, +24 hours
  Nasosorption (vWf antigen)
Circulating inflammatory and oxidative responses after the exposure on the London Underground vs control exposure | -2 hours, +7 hours, +24 hours
  Nasosorption (Thrombin generation)
Circulating inflammatory and oxidative responses after the exposure on the London Underground vs control exposure | -2 hours, +7 hours, +24 hours
  Nasosorption (D-dimer activation)
Circulating inflammatory and oxidative responses after the exposure on the London Underground vs control exposure | -2 hours, +7 hours, +24 hours
  Nasal curettage (mRNA levels to elucidate molecular mechanisms that may explain the toxic effects of particulate matter)
Circulating inflammatory and oxidative responses after the exposure on the London Underground vs control exposure | -2 hours, +24 hours
  Urine (8-isoprostane)
Circulating inflammatory and oxidative responses after the exposure on the London Underground vs control exposure | -2 hours, +24 hours
  Urine (8-hydroxy 2-deoxyguanosine)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Kelly, Principal Investigator — Imperial College London
Locations (1):
- Imperial Clinical Research Facility, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sinharay R, Gong J, Barratt B, Ohman-Strickland P, Ernst S, Kelly FJ, Zhang JJ, Collins P, Cullinan P, Chung KF. Respiratory and cardiovascular responses to walking down a traffic-polluted road compared with walking in a traffic-free area in participants aged 60 years and older with chronic lung or heart disease and age-matched healthy controls: a randomised, crossover study. Lancet. 2018 Jan 27;391(10118):339-349. doi: 10.1016/S0140-6736(17)32643-0. Epub 2017 Dec 5. PMID 29221643